CLINICAL TRIAL: NCT01523366
Title: A Randomized, Open-Label, Multiple Dose, Crossover, Multiple Center Study of the Antiplatelet Effects of Ticagrelor Versus Clopidogrel in Hispanic Patients With Stable Coronary Artery Disease
Brief Title: A Pharmacodynamic Study With Ticagrelor in Hispanic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5130L00012
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Stable Coronary Artery Disease
Keywords: Stable Coronary Artery Disease, CAD
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Min - 90mg/Max - 180mg tablets (loading dose)
  Arms: Ticagrelor
Drug: Clopidogrel — 75mg (once daily)/Max - 600mg tablets (loading dose)
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to assess the pharmacodynamic effect of ticagrelor in Hispanic patients with stable coronary artery disease.

DETAILED DESCRIPTION:
A Randomized, Open-Label, Multiple Dose, Crossover, Multiple Center Study of the Antiplatelet Effects of Ticagrelor versus Clopidogrel in Hispanic Patients with Stable Coronary Artery Disease

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures
* Male or female patients aged 18 years or older Documented stable CAD fulfilling and taking 75-100mg ASA daily treatment
* Females must be post menopausal or surgically sterile Self-identified as Hispanic

Exclusion Criteria:

* Any indication for oral anticoagulant (e.g., atrial fibrillation, mitral stenosis or prosthetic heart valve) or dual antiplatelet treatment (e.g., clopidogrel, prasugrel, ASA dose other than 75 to 100 mg daily) during study period
* Patients who had ACS or stent placed within 12 months of screening Patients with a history of moderate or severe hepatic impairment
* Current smokers, including the use of tobacco containing products in the past 1 month of randomization
* Patients requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Carlson, MD, Study Director — AstraZeneca PharmaceuticalsRoom C3B-718PO Box 15437Wilmington, DE 19850-5437 USA
Locations (5):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Linden, New Jersey

REFERENCES:
- See also: D5130L00012_Clinical_Study_Protocol_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=484&filename=D5130L00012_Clinical_Study_Protocol_Redacted_4-9-14_Redacted.pdf
- See also: CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=484&filename=D5130L00012_CSR_Synopsis_01Apr2014.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from 6 centers in the United States from April 2012 until May 2013.
Pre-assignment Details: 53 patients screened; 40 patients randomized; 38 patients completed the study (7, 8, or 9 days of both treatment sequences), and 39 completed follow-up.
Groups:
- Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence: Ticagrelor 180 milligrams (mg) loading dose followed by 90 mg twice daily (bd) for 7,8 or 9 days (Period 1), and then clopidogrel 600 mg loading dose followed by 75 mg once daily (od) for 7, 8 or 9 days (Period 2).
- Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence: Clopidogrel 600 mg loading dose followed by 75 mg od for 7, 8 or 9 days (Period 1), then ticagrelor 180 mg loading dose followed by 90 mg bd for 7,8 or 9 days (Period 2)
Period: Treatment Period 1
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout Period - 10-14 Days
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence
Started | 19 | 20
Completed | 18 | 20
Not Completed | 1 | 0
Not completed — Not completed at least 7 days treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set for demography (N=40) - included all patients who signed informed consent and were randomized into the study. Pharmacodynamic (PD) Analysis Set for outcomes (N=38) - included all patients for whom PD data was available with no major protocol deviations thought to significantly affect the PD of ticagrelor or clopidogrel
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 10 | 8 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 17 | 18 | 35
  Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 20 | 20 | 40
  Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 20 | 40
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of the P2Y12 Receptor as Measured by P2Y12 Reactions Units (PRU) From VerifyNow™ (a Platelet Function Test Developed by Accumetrics) at 2 Hours After Loading Dose
Description: Participants with low (<150) baseline PRU values (indicating an incomplete washout from anti-platelet therapy) were excluded during the period corresponding to the low baseline value
Time Frame: At 2 hours after the loading dose
Population: Pharmacodynamic (PD) Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Groups:
- Ticagrelor Arm: Ticagrelor 180 mg loading dose followed by 90 mg bd for 7,8 or 9 days.
- Clopidogrel Arm: Clopidogrel 600 mg loading dose followed by 75 mg od for 7, 8 or 9 days.
Arm/Group | Ticagrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 37 | 34
PRU | 34.2 [12.4 to 55.9] | 201.4 [178.7 to 224.1]
Statistical Analysis 1: Comparison: Ticagrelor Arm vs Clopidogrel Arm; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Model contained treatment group, period, and sequence as fixed effects, and a random effect for participant within sequence; Mean Difference (Final Values) = -167.2, 95% CI 2-sided [-197.0 to -137.4], Standard Error of Mean 14.6 — Ticagrelor minus clopidogrel

2. Secondary Outcome: Inhibition of the P2Y12 Receptor as Measured by PRU From VerifyNow™ at 0.5 and 8 Hours After Loading Dose
Description: as for outcome 1
Time Frame: At 0.5 and 8 hours after the loading dose
Population: PD Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Arm/Group | Ticagrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 38 | 34
PRU
  0.5 hours | 134.6 [105.1 to 164.1] | 269.8 [238.7 to 300.8]
  8 hours | 34.0 [9.2 to 58.8] | 202.8 [176.6 to 229.0]
Statistical Analysis 1: Comparison: Ticagrelor Arm vs Clopidogrel Arm; Analysis at 0.5 hours after the loading dose; Test type: Superiority or Other; p < .001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -135.2, 95% CI 2-sided [-172.3 to -98.0], Standard Error of Mean 18.23 — Ticagrelor minus Clopidogrel
Statistical Analysis 2: Comparison: Ticagrelor Arm vs Clopidogrel Arm; Analysis at 8 hours after the loading dose; Test type: Superiority or Other; p < .001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -168.9, 95% CI 2-sided [-204.0 to -133.7], Standard Error of Mean 17.28 — Ticagrelor minus Clopidogrel

3. Secondary Outcome: Inhibition of the P2Y12 Receptor as Measured by PRU From VerifyNow™ at 2 and 8 Hours on Day 7 After Multiple Doses and at End of Dosing Interval on Day 8
Description: The end of dosing interval was approximately 12 hours after the last evening dose of ticagrelor and approximately 24 hours after the last morning dose of clopidogrel. Participants with low (<150) baseline PRU values (indicating an incomplete washout from anti-platelet therapy) were excluded during the period corresponding to the low baseline value
Time Frame: At 2 hours and 8 hours on Day 7 after multiple doses, and at the end of dosing interval on Day 8
Population: PD Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Arm/Group | Ticagrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 37 | 34
PRU
  2 hours on day 7 | 28.5 [8.0 to 49.0] | 179.0 [157.7 to 200.3]
  8 hours on Day 7 -ticagrelor N=36 clopidogrel N=33 | 38.7 [17.2 to 60.3] | 178.9 [156.5 to 201.4]
  End of Dosing Interval on Day 8 - N's per 8 hours | 51.5 [29.8 to 73.1] | 182.1 [159.5 to 204.7]
Statistical Analysis 1: Comparison: Ticagrelor Arm vs Clopidogrel Arm; Analysis at 2 hours on Day 7 after multiple doses; Test type: Superiority or Other; p < .001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -150.5, 95% CI 2-sided [-176.9 to -124.1], Standard Error of Mean 12.97 — Ticagrelor minus Clopidogrel
Statistical Analysis 2: Comparison: Ticagrelor Arm vs Clopidogrel Arm; Analysis at 8 hours on Day 7 after multiple doses; Test type: Superiority or Other; p < .001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -140.2, 95% CI 2-sided [-168.4 to -111.9], Standard Error of Mean 13.84 — Ticagrelor minus clopidogrel
Statistical Analysis 3: Comparison: Ticagrelor Arm vs Clopidogrel Arm; Analysis at end of dosing interval on Day 8; Test type: Superiority or Other; p < .001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -130.6, 95% CI 2-sided [-158.0 to -103.2], Standard Error of Mean 13.41 — Ticagrelor minus clopidogrel

4. Secondary Outcome: Ticagrelor Plasma Concentrations After the Loading and Maintenance Doses
Description: The standard deviation (SD) is a statistic using the log-transformed data and is not the geometric SD.
Time Frame: Predose, 0.5, 2, 8 hours from loading dose; 0, 2, 8 and 12 hours from last dose
Population: Pharmacokinetic (PK) Analysis Set, defined as all participants for whom at least one valid PK reading was available
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Ticagrelor (Treatment Period 1); Ticagrelor (Treatment Period 2): Ticagrelor 180 mg loading dose followed by 90 mg bd for 7, 8 or 9 days
Arm/Group | Ticagrelor (Treatment Period 1) | Ticagrelor (Treatment Period 2)
Number analyzed (Participants) | 18 | 19
ng/mL
  Baseline (0 hours - pre-dose) | 1.2 (7.5) | 1.1 (1.8)
  0,.5 hours after the loading dose | 206.7 (413.1) | 118.6 (352.0)
  2 hours after the loading dose - Period 2 N=18 | 665.4 (566.2) | 758.5 (716.6)
  8 hours after the loading dose | 376.9 (378.8) | 479.6 (210.7)
  0 hours after multiple doses | 248.8 (238.9) | 220.1 (295.8)
  2 hours after multiple doses | 609.3 (271.3) | 466.5 (534.5)
  8 hours after multiple doses | 340.4 (283.8) | 305.2 (301.6)
  End of dosing interval on Day 8 - Period 1 N=17 | 283.3 (438.1) | 200.7 (268.4)

5. Secondary Outcome: AR-C124910XX (an Active Metabolite of Ticagrelor) Plasma Concentrations After the Loading and Maintenance Doses
Description: The SD is a statistic using the log-transformed data and is not the geometric SD.
Time Frame: Predose, 0.5, 2, 8 hours from loading dose; 0, 2, 8 and 12 hours from last dose
Population: PK Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor (Treatment Period 1) | Ticagrelor (Treatment Period 2)
Number analyzed (Participants) | 18 | 19
ng/mL
  Baseline (0 hours - pre-dose) | 1.1 (2.3) | 1.0 (0.0)
  0,.5 hours after the loading dose | 13.6 (66.3) | 9.3 (26.9)
  2 hours after the loading dose - Period 2 N=18 | 153.2 (128.6) | 170.8 (156.5)
  8 hours after the loading dose | 113.8 (54.6) | 97.7 (61.9)
  0 hours after multiple doses | 113.3 (102.1) | 62.7 (76.7)
  2 hours after multiple doses | 183.4 (120.8) | 97.4 (147.9)
  8 hours after multiple doses | 132.8 (61.9) | 83.5 (71.4)
  End of dosing interval on Day 8 - Period 1 N=17 | 124.8 (56.6) | 57.7 (83.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signature of the informed consent throughout the treatment period including the follow up visit (approximately 11 weeks for each participant).
Description: Adverse events were solicited at each scheduled visit and could be reported by the participant at any time during the study. When summarizing Treatment Period 1 and Treatment Period 2 totals, each participant was counted only once for an individual adverse event, regardless of whether it occurred on ticagrelor, clopidogrel or both.
Arm/Group | Ticagrelor Arm | Clopidogrel Arm
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 5/40 | 6/39
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor Arm (N=40) | Clopidogrel Arm (N=39)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Burning Sensation (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Total N for the secondary outcome analysis after multiple doses and for PK measures was not the same for 2 hours, 8 hours and end of dosing. Only the first time point total N can be reported via the form. Row titles indicate N's where they differ.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AstraZeneca (AZ) for review at least 60 days in advance of the submission for publication. The Investigators in the Multi-Center (MC) study agree to postpone MC publications until the earlier of the first AZ-authorized publication or up to 18 months from study completion at all sites.